CLINICAL TRIAL: NCT06007196
Title: Performance Evaluation of Non-invasive Continuous Hemodynamic Measurement From Task Force(R) CORE Versus Invasive Reference
Brief Title: Evaluation of Non-invasive Continuous Hemodynamic Measurement From Task Force CORE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Christian Reiterer, Principal Investigator, Medical University of Vienna
Other Study IDs: Task_Force_01
Record Dates: First submitted 2023-07-07; First posted 2023-08-23 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Hemodynamic Measurement; Non-invasive; Cardiac Output

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Continuous non-invasive Hemodynamic Monitoring: Continuous non-invasive Hemodynamic Monitoring (Task Force CORE(R) and Task Force CARDIO(R)) will be compared to invasive thermodilution cardiac output measurements in all patients.
  Interventions: Device: non-invasive device (Task Force CORE(R) and Task Force CARDIO(R)

INTERVENTIONS:
Device: non-invasive device (Task Force CORE(R) and Task Force CARDIO(R) — Intraoperative cardiac output will be measured using the non-invasive device (Task Force CORE(R) and Task Force CARDIO(R) and will be compared with the invasive thermodilution method (PiCCO).

SUMMARY:
Validation of hemodynamic measurements using the non-invasive Task Force Core(R) and Task Force Cardio(R) device with invasive hemodynamic measurements using the thermodilution technique (PICCO device).

DETAILED DESCRIPTION:
The investigational device, Task Force® CORE (TFC, CNSystems Medizintechnik GmbH, Graz, Austria) together with the Task Force® CARDIO (TFCARDIO, CNSystems Medizintechnik GmbH, Graz, Austria) medical device software, is a new CE-marked medical device for continuous non-invasive determination of blood pressure (BP), cardiac output (CO) and derived parameters based on the well established CNAP® (continuous non-invasive arterial pressure) technology by CNSystems. The primary aim of this prospective, method comparison, open, multi-center study is data acquisition for the performance evaluation of the TFC in comparison with invasive reference methods (i.e. transpulmonary thermodilution, invasive blood pressure with radial artery catheter). The setting of the study will be the Operating Room (OR). This setting allows the comparison of the investigational device's cardiac output (CO) to invasive CO as well as of BP and derived hemodynamic parameters like Stroke Volume (SV), and Systemic Vascular Resistance (SVR). Measurements will be performed during the perioperative period, starting 15 minutes after the first skin incision.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (patients aged at least 18 years)
* Patients undergoing major abdominal surgery who require invasive extended hemodynamic monitoring (trans pulmonary thermodilution via PiCCO and invasive blood pressure monitoring with radial artery catheter) according to clinical standard of care
* Patients with intact perfusion of both hands evidenced by a positive Allen's test
* Patients given written informed consent to participate in the study

Exclusion Criteria:

* Patients with vascular impairments at the sites of non-invasive blood pressure measurement (fingers or upper arms)
* Patients with significant edema in the fingers
* Patients with ventricular assist devices or extracorporeal life-supporting devices
* Subjects not passing the Allen's test for both hands
* Patients who obtain vasoactive medications on the same arm as used for upper-arm Task Force blood pressure measurements
* Patients with a large lateral difference in blood pressure (> 15mmHg for systolic blood pressure and/or >10 mmHg for diastolic blood pressure) or with same arm measurement differences > 10 mmHg in systolic or diastolic blood pressure during assessment of lateral differences
* Patients who, in addition to invasive blood pressure monitoring, require non-invasive blood pressure measurements unrelated to the investigational device

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients, who undergo major abdominal surgery, which will require extended hemodynamic monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference in intraoperative cardiac output measurements between Task Force CORE compared with thermodilution during surgery | For the duration of surgery
  Intraoperative performance of cardiac output values derived by the Task Force CORE system compared with cardiac output measurements derived by thermodilution measurements.

SECONDARY OUTCOMES:
Differences in intraoperative hemodynamic measurements (blood pressure in mmHg) between Task Force CORE compared with thermodilution during surgery | For the duration of surgery
  Intraoperative evaluation of the performance of Task Force variable blood pressure (in mmHg) throughout surgery compared to simultaneous invasive measurements.
Differences in intraoperative hemodynamic measurements (stroke volume in ml) between Task Force CORE compared with thermodilution during surgery | For the duration of surgery
  Intraoperative evaluation of the performance of Task Force variable stroke volume (in ml) throughout surgery compared to simultaneous invasive measurements.
Differences in intraoperative hemodynamic measurements (stroke volume variation in %) between Task Force CORE compared with thermodilution during surgery | For the duration of surgery
  Intraoperative evaluation of the performance of Task Force variable stroke volume variation (in %) throughout surgery compared to simultaneous invasive measurements.
Intraoperative continuous Cardioc Output measurements | For the duration of surgery
  The comparison of intraoperative continuous cardiac output measurements derived by the Task Force device with continuous invasive cardiac output measurements derived by the PiCCO throughout surgery or before, during and after clinically indicated interventions (e.g. medication, passive leg raising, fluid challenge).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria